CLINICAL TRIAL: NCT00976482
Title: Clinical Outcome of Pacemaker paTIents According to Pacing Modality and Primary INDications
Acronym: OPTI-MIND
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-09
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Bradyarrhythmia
Keywords: Cardiovascular; Pacemaker; Mortality; Physiologic pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker: Patients currently implanted with permanent Pacemaker according to guidelines

SUMMARY:
The study objective is to collect mid-term clinical outcome in a group of patients implanted with permanent pacemaker (PM) according to real-life clinical practice in a multicenter and international environment.

DETAILED DESCRIPTION:
The principal objective of the OPTI-MIND study is to collect data on two-year all-cause mortality in a general population implanted with a PM according to current clinical practice. Additionally, the study aims to stratify the outcome by both known patient-related risk factors and by physiologic pacing mode setting (a specifically defined PM programming). Stratification will be done for pre-specified classes of patients on the basis of their primary rhythm disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a current Boston Scientific pacemaker (all ALTRUA models) or any future commercially available Boston Scientific PM families according to international and local guidelines for pacemaker implantation;
* Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational centre;
* Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Unable to be followed up by the participating centres for a period of two years;
* Current device implanted for more than 15 days;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry or extensions/amendments of the current protocol. Each instance should be brought to the attention of the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with permanent pacemaker accroding to guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1745 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Biffi, MD, Study Chair — Az. Osp. S. orsola - Malpighi, Bologna, Italy
Locations (1):
- Katholisches Krankenhaus, St.Johannes Hospital, Hagen, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacemaker
Started | 1745
Eligible for Last Follow up | 1487
Completed | 1486
Not Completed | 259
Not completed — Death | 208
Not completed — Withdrawal by Subject | 45
Not completed — Center terminated | 1
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: among the 1745 initial patients 5 were excluded for inclusion criteria violations (deviations from correct signature of informed consent)
Arm/Group | Pacemaker
Number analyzed (Participants) | 1740
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (10)
Gender [Count of Participants; unit: Participants]
  Female | 1047
  Male | 693
Primary Indication for Permanent Pacing [Number; unit: participants]
  sinus node dysfunction | 565
  Atrioventricular Block | 840
  Neuro-mediated | 61
  Permanent AF with Slow Ventr. Response | 274

OUTCOME MEASURES:

1. Primary Outcome: Two-year All-cause Mortality
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker
Number analyzed (Participants) | 1740
percentage of participants | 11 [9.3 to 13.8]

ADVERSE EVENTS:
Groups:
- Pacemaker: implanted Patients
Arm/Group | Pacemaker
Serious Adverse Events (participants affected / at risk) | 611/1740
Other Adverse Events (participants affected / at risk) | 206/1740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker (N=1740)
disease progression leading to death (Cardiac disorders) | 208 (208)
leading to invasive interventions (Cardiac disorders) | 403 (632)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacemaker (N=1740)
atrial fibrillation (Cardiac disorders) | 206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days